CLINICAL TRIAL: NCT06901232
Title: Effect of Network-based Real Time Neurofeedback Augmentation of Mindfulness Practice on Recurrent Negative Thinking in Adolescents at Risk for Serious Mental Illness
Brief Title: Mindfulness-based Neurofeedback to Reduce Negative Thinking in CHARMS Adolescents
Acronym: CHARMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Anne Eden Evins, Founding Director Massachusetts General Hospital Center for Addiction Medicine; Cox Family Professor of Psychiatry, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2024P003611
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Repetitive Negative Thinking; Serious Mental Illness Symptoms
Keywords: Mindfulness; Repetitive negative thinking; Serious mental illness symptoms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active mindfulness-based neurofeedback (Active mbNF) (Experimental): Participants will:
  * Receive a 45-minute mindfulness training
  * Receive two sessions of active mindfulness-based neurofeedback
  Interventions: Behavioral: Mindfulness Training; Behavioral: Active mindfulness-based neurofeedback (Active mbNF)
- Sham mindfulness-based neurofeedback (Sham mbNF) (Sham Comparator): Participants will:
  * Receive a 45-minute mindfulness training
  * Receive two sessions of sham neurofeedback
  Interventions: Behavioral: Mindfulness Training; Behavioral: Sham mindfulness-based neurofeedback

INTERVENTIONS:
Behavioral: Mindfulness Training — All participants will complete a single 45-minute mindfulness training at Visit 2, with a refresher prior to the second mbNF session at Visit 3. Clinically trained study staff will conduct the training with the aim of teaching "mental noting," a core mindfulness technique to be practiced and employed during neurofeedback. Mental noting is a major component of Vipassana (insight mindfulness meditation); its key principles include: "concentration", "observing sensory experience,'' "not 'efforting'", and "contentment".Specifically, participants will be taught to mentally label/note whatever sensation is most prominent in their sensory experience from moment to moment (e.g., seeing, hearing, feeling, thinking). Training will be personalized to identify scenarios in which mental noting can be applied in the context of each person's daily life, explaining the goal of using these strategies to manage distress in daily life.
Behavioral: Active mindfulness-based neurofeedback (Active mbNF) — Before the MRI scan, participants will practice mental noting by verbalizing their mental label with the study clinician providing feedback. Participants will then complete a silent practice of mental noting while viewing simulated neurofeedback. Participants will be trained until they feel competent to use mental noting in the scanner. During active mbNF (6 runs, 2.5 minutes each), participants will use mental noting with the aim of controlling visual feedback. Specifically, they will attempt to move the position of the white dot toward the (upper) red circle and away from the (lower) blue circle.
  Arms: Active mindfulness-based neurofeedback (Active mbNF)
Behavioral: Sham mindfulness-based neurofeedback — Before the MRI scan, participants will practice mental noting by verbalizing their mental label with the study clinician providing feedback. Participants will then complete a silent practice of mental noting while viewing simulated neurofeedback. Participants will be trained until they feel competent to use mental noting in the scanner. During sham mbNF, participants will view a visual display (white dot, red and blue circles) extracted from a previously acquired mbNF session. The display will be independent from brain activity in the sham condition and will simply mirror the stimuli observed by those in the mbNF group. This ensures participants across groups are viewing equivalent stimuli for the same amount of overall time.
  Arms: Sham mindfulness-based neurofeedback (Sham mbNF)

SUMMARY:
The study will test the hypothesis that mindfulness-based neurofeedback (mbNF) will improve repetitive negative thinking and social and role functioning over sham neurofeedback in adolescents at risk for serious mental illness. To do so, 90 adolescents ages 14-21 with elevated repetitive negative thinking will be enrolled into a double-blind randomized clinical trial of sessions of mindfulness training with either active mindfulness-based neurofeedback or sham neurofeedback and three months of mindfulness practice and follow up.

DETAILED DESCRIPTION:
Approximately 90 at-risk adolescents ages 14-21 years old will be enrolled in a double-blind, randomized clinical trial. All participants will undergo a baseline clinical assessment (Visit 1), which will serve as an important baseline for daily symptom fluctuation and use of mindfulness strategies prior to training. Approximately 1-2 weeks after the baseline assessments, all participants will complete an in-person visit (Visit 2) in which they will complete a brief MRI scan (resting state localizer) and a 45-minute mindfulness training. After the mindfulness training, participants will be randomized in a 1:1 ratio to receive either active or sham neurofeedback (n=45 each group). Randomization will be stratified by information obtained at the baseline assessment: biological sex, prior daily/near daily mindfulness practice for 8 weeks or more. A study staff member with no participant contact will create randomization tables in REDCap to alloacte participants to either active or sham mbNF. Participants and staff will remain blinded to assignment. Participants will then complete another MRI session what will include resting state scans as well as the active or sham mbNF. Approximately 1-2 weeks later, participants will return for another in-person visit (Visit 3) that includes a mindfulness refresher and repeats the procedures of Visit 2. Participants will briefly rate their mindfulness practice daily for three months using a brief, online survey. At 1-, 3- and 12-months post-neurofeedback, participants will complete self-report and clinician-rated assessments to probe repetitive negative thinking and prodromal psychiatric symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Ages 14-21, inclusive
* Recurrent negative thinking, defined as PTQ-C (<18 years) or PTQ (18 years or older) total score >30 and at least two questions scored 3 or 4.
* Able to understand study procedures, read, and write in English
* If age is 18 years or older: Competent and willing to provide written informed consent
* If age is less than 18 years: Competent and willing to provide written informed assent AND have a parent/legal guardian who is competent and willing to provide written informed consent
* Access to a mobile device to complete daily survey assessments

Exclusion Criteria:

* Any of the following lifetime mental health disorders by DSM-V criteria: psychotic disorders, anxiety disorder, bipolar disorder, oppositional defiant disorder, conduct disorder, developmental disorder (e.g., autism), post-traumatic stress disorder, or eating disorder
* Substance use disorder, moderate or severe in past six months.
* Unstable medical or neurologic condition, epilepsy or seizure disorder, head injury, loss of consciousness >5 minutes
* MRI contraindications (i.e. presence of ferromagnetic implants, cardiac pacemaker or pacemaker wires, metallic particles in the body, vascular clips in the head or previous neurosurgery, prosthetic heart valves, magnetic dental implants claustrophobia).
* Visual, auditory, or cognitive impairment (IQ<80 based on the Wechsler Abbreviated Intelligence Scale (WASI)) that may make it difficult to participate.
* Any condition or situation that would, in the investigator's opinion, make it unlikely that the participant could adhere safely to the study protocol.
* Pregnancy; a negative pregnancy test is required at enrollment
* Individuals who are under the legal protection of the government or state (Wards of the State)
* Inability to speak, read, or write English fluently

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2027-09 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Change in repetitive negative thinking (RNT) | 2 weeks
  Perseverative Thinking Questionnaire- Child Version (PTQ-C), is a content-independent measure of RNT, with 15 items, rated on a 5- point scale (never, almost never, sometimes, often, almost always), with excellent internal consistency, Cronbach's alpha=0.95, in both clinical and non-clinical samples, validated and normed in clinical and non-clinical adolescent and young adult samples as a transdiagnostic research tool that has been shown to predict MDD. Higher scores indicate greater RNT.

SECONDARY OUTCOMES:
Change in psychotic symptom severity | 2 weeks
  Psychotic symptoms will be assessed using the Brief Psychiatric Rating Scale (BPRS), a well validated, 18-item, interview-based measure of positive and negative psychotic, depressive, and general psychiatric symptoms that is sensitive to treatment effects and is included in the PhenXToolkit. Scores for each item range from 1 (not present) and 7 (extremely severe). Higher scores indicate greater severity of psychotic symptoms.
Change in depressive symptom severity | 2 weeks
  Depressive symptoms will be assessed by the Quick Inventory of Depressive Symptoms - (QIDS-C) for participants ages 18 and older and the Quick Inventory of Depressive Symptoms - Adolescent Version (QIDS-A17) for participants under 18 years old. The QIDS is a 17-item clinician rated scale that assesses mood, sleep, appetite, and suicidal ideation. Higher scores indicate greater depressive symptom severity.
Change in social and occupational functioning | 2 weeks
  Social and occupational functioning will be assessed using the Social and Occupational Functioning Assessment Scale (SOFAS). It focuses exclusively on the individual's level of social and occupational functioning and is not directly influenced by the overall severity of the individual's psychological symptoms. Scores range from 0 to 100, with lower scores indicating greater levels of impairment.
Change in worry symptom severity | 2 weeks
  The Penn State Worry Questionnaire will be used to assess RNT in the form of worry. The scale has a possible range from 0 to 42. Severity cutoffs are as follows: normal (0-15), at risk (top 3-7%; 16-18), clinically elevated (top 2%; 19+). Participants under 18 years old will be assessed using the Penn State Worry Questionnaire for Children.
Change in rumination symptom severity | 2 weeks
  The Rumination Response Scale (RRS) will be used to assess RNT in the form of depressive content and response styles for depression. The scale is 22 items and each item is rated on a 4-point Likert scale, with responses ranging from 1 (almost never) to 4 (almost always). Higher scores indicate more severe rumination responses.

CONTACTS AND LOCATIONS:
Overall Officials: A. Eden Evins, MD, MPH, Principal Investigator — Massachusetts General Hospital; Susan Whitfield-Gabrieli, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Center for Addiction Medicine, 101 Merrimac Street, Suite 320, Boston, MA 02114, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available upon request. Data will include de-identified individual patient-level data and a data dictionary. Investigators proposing to use the data must execute a data use agreement with Massachusetts General Hospital and have approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, before data is shared. Data will be available within three months of manuscript publication. Requests for data should be sent to aeevins@mgh.harvard.edu.
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following manuscript publication.